CLINICAL TRIAL: NCT03877289
Title: Efficacy of Oxybutynin in Paediatric Cystitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, David W Johnson, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: OxyRCT1
Record Dates: First submitted 2019-01-16; First posted 2019-03-15 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Cystitis
Keywords: pediatrics; cystitis; UTI; oxybutynin
MeSH Terms: conditions — Cystitis | interventions — oxybutynin; Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxybutynin (Experimental): Children aged 4 - 6 years: Oxybutynin 2.5 mg (2.5ml) po TID Children aged 7 - 16 years: Oxybutynin 5 mg (5ml) po TID
  Interventions: Drug: Oxybutynin; Drug: Antibiotics
- Placebo (Placebo Comparator): Orasweet liquid placebo
  Interventions: Other: "Orasweet" Liquid Placebo; Drug: Antibiotics

INTERVENTIONS:
Drug: Oxybutynin — Oxybutynin is a tertiary amine anticholinergic. It exerts both antispasmodic and antimuscarinic activity on smooth muscle. It also exerts analgesic and local anaesthetic effects.
  Arms: Oxybutynin
Other: "Orasweet" Liquid Placebo — A formulated Oxybutynin placebo that is nearly identical in appearance, volume, weight, taste, and smell.
  Arms: Placebo
Drug: Antibiotics — All patients in treatment and control arms were treated as a co-intervention with an oral antibioitic, the type of which was chosen by the child's attending physician.
  Possible prescribed antibiotics include: trimethoprim and sulfamethoxazole (Septra), Cefalotin, Cephalexin, Cefapirin, Cefdroxil, Cefazolin, Cefradine, Cefacetrile, Cefaloridine, Cefroxadine, Cefatrizine, Cefuroxime, Cefixime, amoxicillin/clavulanic acid (Clavulin), and Nitrofurantoin.

SUMMARY:
The primary goal of this study is to determine if the addition of the bladder antispasmotic oxybutynin to standard antimicrobial therapy in the treatment of childhood cystitis will decrease the associated pain and discomfort. A randomized, double blind, placebo-controlled clinical trial design will be used. The second goal of this study will be to describe the nature and duration of symptoms associated with uncomplicated cystitis in the paediatric age group. Finally, adverse side effects associated with short term use of oxybutynin will be monitored.

DETAILED DESCRIPTION:
Roughly half of children age 4 to 16 who are diagnosed with a UTI have cystitis. Adult sufferers of cystitis report terrible scorching with voiding, frequent sensation of the need to void with little results, and aching and pressure in the abdomen and genitals. The management of cystitis in adulthood often includes medication directed at easing pain and discomfort. Little research has been directed at documenting the true incidence of these unpleasant symptoms in paediatric cystitis and virtually no literature exists on the management of the associated pain and discomfort. This study will aim to describe the nature and duration of unpleasant symptoms suffered by children with cystitis and will investigate the efficacy of a possible therapy to ease their suffering.

Hypothesis: The investigators feel that oxybutynin is the most suitable agent for the first trial of bladder antispasmodics in paediatric cystitis. The investigators reasoning is as follows:

1. Previous adult studies have favored an anticholinergic agent (flavoxate) over the topical analgesic phenazopyridine in the symptomatic treatment of cystitis.
2. Newer anticholinergic agents such as oxybutynin and tolterodine have been shown to be superior to older anticholinergic agents (such as flavoxate) in the treatment of many uncomfortable conditions of the bladder.
3. Oxybutynin has been extensively studied in children for several non-infectious conditions of the bladder. The safety profile, expected side effects and dosage range have therefore been established for children.
4. Oxybutynin is marketed in a palatable syrup. A placebo can easily be manufactured that is identical in taste, texture, smell, color, and volume.

The study will be a randomized, double-blind, placebo controlled clinical trial of oxybutynin therapy for symptom control in paediatric cystitis. Toilet trained children aged 4 - 16 years who present to the Alberta Children's Hospital (ACH) emergency room and receive a diagnosis of cystitis are eligible to participate.

ELIGIBILITY:
Inclusion Criteria:

1. Age 4 - 16 years
2. Suspected diagnosis of cystitis based on a clean catch or catheter urinalysis (must have at least one of the three screening tests positive - leukocyte esterase, nitrites, or leukocytosis or bactiuria on microscopy)
3. Intention to manage patient as an out-patient with oral antibiotics
4. Parent must be available to assist younger children with the measurements for 24 hours and must be willing to receive follow-up calls daily until symptoms resolve
5. Written informed consent (and assent when age-appropriate)

Exclusion Criteria:

1. Clinically suspected pyelonephritis (ED temperature > 38.5, significant flank pain, vomiting > 3 times/24 hours)
2. Patient not toilet trained
3. Patient with significant language delays (preventing use of the facial pain scale)
4. Patient with sensory deficits at the sacral level
5. Inability of the patient and parent to speak and understand English
6. Known contraindication to Oxybutynin (hypersensitivity, glaucoma, bowel obstruction, megacolon, ulcerative colitis, myesthenia gravis, renal or hepatic disease, hyperthyroidism, heart disease, and obstructive uropathy)
7. Patient on any medications during the preceding 8 hours that have analgesic or anticholinergic properties (acetominophen, and inhaled medications will be permitted)
8. Patients who have been previously enrolled in the study
9. Lack of a telephone in the home
10. Known or suspected pregnancy or lactation in the patient
11. Treating physician uses pyridium

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2008-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Pain/discomfort ratings obtained at 4 hours after each of the three doses of study medication. | Four hours after each of the three doses of study medication.
  Participants will be asked to rate how they feel at each of these times using the McGrath Facial Affective Scale (MFAS). The MFAS ranges from the lowest pain score A (happy face) to the highest pain score I (very unhappy crying face). Data will be acquired over a 4 hours after the oxybutynin is given, therefore the investigators can expect that some of the measurements will be disrupted by nighttime sleep for some of the participants. Parents will be asked to document if their child is sleeping during the time when measurements are to be made.

SECONDARY OUTCOMES:
Measurements of pain/discomfort with each urination recorded during the first 24 hours. | Immediate 24 hours after presenting to the ED.
  Measurements will be made using the McGrath Facial Affective Scale and will be recorded by the participant or family member at home.
Number of supplemental doses of acetominophen used during the first 24 hours of the study. | Immediate 24 hours after presenting to the ED.
  This information will be recorded by the participant or caregiver at home.

CONTACTS AND LOCATIONS:
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No